CLINICAL TRIAL: NCT03715192
Title: Single-Ascending Dose, Safety, Tolerability, and Pharmacokinetic Study of LY3462817
Brief Title: A Safety Study of LY3462817 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17089; J1A-MC-KDAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3462817 - IV (Experimental): Escalating doses of LY3462817 administered as a single intravenous (IV) infusion in healthy participants
  Interventions: Biological: LY3462817 IV
- Placebo (Placebo Comparator): Normal saline administered as a single IV infusion in healthy participants
  Interventions: Drug: Placebo
- LY3462817 - SC (Experimental): Single dose of LY3462817 administered as subcutaneous (SC) injections in healthy participants
  Interventions: Biological: LY3462817 SC

INTERVENTIONS:
Biological: LY3462817 IV — Administered IV
  Arms: LY3462817 - IV
Biological: LY3462817 SC — Administered SC
  Arms: LY3462817 - SC
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
This study is being conducted to determine how safe and how well tolerated LY3462817 is when given intravenously (IV) (into a vein) and subcutaneously (SC) (just under the skin) to healthy participants. Blood tests will be done to check how much LY3462817 is in the bloodstream and how long the body takes to get rid of it. Each enrolled participant will receive 1 dose of LY3462817 or placebo. The study will last about 16 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female who cannot get pregnant
* Have a body mass index (BMI) of 18 to 32 kilogram per square meter (kg/m²), inclusive, at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG, heart tracing), blood and urine laboratory test results that are acceptable for the study
* Weight at least 45 kilograms (kg)

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have cancer or a malignant disease in the past 5 years
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Are unwilling to receive study drug administration by injections or through the veins

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | Baseline through to final follow-up at approximately Week 12
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) of LY3462817 | Baseline through to final follow-up at approximately Week 12
  Pharmacokinetics: Cmax of LY3462817
Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) of LY3462817 | Baseline through to final follow-up at approximately Week 12
  Pharmacokinetics: AUC of LY3462817

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Nus Centre for Clin Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No